CLINICAL TRIAL: NCT02014597
Title: Use of a Novel, Objective Optokinetic Contrast Device to Determine Scotopic Range Visual Function and Discriminate Between Patients With and Without Glaucoma
Brief Title: Human Optokinetic Contrast Device (HOCD) to Measure Visual Function and Identify Patients With and Without Glaucoma
Acronym: HOCD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding lapse; enrollment difficulty
Sponsor: Benjamin Frankfort, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Benjamin Frankfort, MD, PhD, Associate Professor, Principal Investigator, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-30109
Record Dates: First submitted 2013-11-26; First posted 2013-12-18 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Normal - No glaucoma (Experimental): HOCD
  Interventions: Device: HOCD
- Glaucoma (Experimental): HOCD
  Interventions: Device: HOCD

INTERVENTIONS:
Device: HOCD — feasibility of HOCD and comparison of HOCD results between subjects with and without glaucoma

SUMMARY:
The purpose of this study is to determine if an optokinetic contrast detection device is sufficient to measure contrast sensitivity and to distinguish between patients with and without glaucoma.

DETAILED DESCRIPTION:
The protocol is divided into two studies that will have two separate consent forms (Study 1 and Study 2).

Study 1 involves the optimization of the device parameters. Study 1 will test adult subjects with no history of ocular disease (Study 1A) to assess the limits of human contrast sensitivity and subjects with definite glaucoma (Study 1B) by gathering preliminary data for comparison. These two pilot sub-studies intend to provide rapid data in regard to the device testing results to support the study hypothesis. This strategy will help rule out false negatives and false positives so that any adjustments can be made prior to the start of Study 2 for longitudinal data collection. Study 2 involves determination of baseline population parameters for an older population more likely to be age-matched with patients with glaucoma, as well as performance of patients with various levels of glaucoma severity.

Enrollment of participants in Study 1B will begin after the first 5 participants have been enrolled and tested in Study 1A. Study 2 will begin after Study 1A and B are complete.

Study 1: No more than 20 adult subjects with no history of ocular disease and no more than 20 adults subjects with definite glaucoma will be recruited to assist with optimization of device parameters.

Study 1A: The individuals will not be patients of the co-investigators but rather volunteers who are recruited by word of mouth (co-employees, residents, research staff, etc.) and are willing to volunteer their time to assist in the development of the project. Volunteers can be of any age >18, male or female, and must be of self-reported excellent ocular health. Best spectacle corrected visual acuity of 20/40 or better is required (verified by Snellen acuity testing on the day of participation) and the participant must have no reported history of glaucoma, retinal disease, amblyopia, ocular trauma, or ocular surgery of any kind with the exception of refractive surgery (LASIK, PRK, or equivalent).

Study 1B: These individuals will be recruited from the Alkek Eye Center patient population with confirmed diagnosis of glaucoma and of any age > 18.

Study 2: Potential subjects will be recruited from the Department of Ophthalmology at Baylor College of Medicine and their families. We will recruit 100 patients for this study in the following distribution:

1. 20 normal controls age 50 or older
2. 20 patients age 50 or older with ocular hypertension
3. 20 patients age 50 or older who are glaucoma suspects
4. 20 patients age 50 or older with early to moderate glaucoma
5. 20 patients age 50 or older with moderate to advanced glaucoma

Study 1: Subjects participating in this portion of the study will attend one single visit: 1) Informed consent will be obtained and inclusion/exclusion criteria will be confirmed. Demographic information, ocular history, refraction, and visual acuity information will be collected for all patients. Additional clinical data will also be collected for Study 1B participants only. Information to be collected will include name, date of birth, ethnicity, gender, ocular history (surgery, etc), type of glaucoma (Study 1B), current visual acuity, refraction, central corneal thickness (Study 1B), intraocular pressure (Study 1B), recent slit lamp exam including lens status (Study 1B), recent dilated exam including optic nerve appearance (Study 1B), and recent automated perimetry results (Humphrey visual field, Study 1B) 2) Snellen visual acuity will be measured while wearing current spectacle correction to ensure acuity of 20/40 or better. The current spectacle correction (refraction) and acuity will be recorded. 3) OKR (optokinetic reflex)-based contrast testing will be performed with the OCD - optokinetic contrast device (the device in study with this protocol). Subjects will be shown a brief demonstration of the OCD under red light (to begin dark adaptation) to familiarize themselves with the device and the expected testing strategy. 4) Subjects will then be dark adapted for 20-30 minutes. During this time they will be sitting in a darkened room. If the room is not dark enough a loose blindfold may be used. Music options will be available to help pass the time and ease potential discomfort. 5) After 20-30 minutes the blindfold will be removed (if used) and patient will have monocular dark-adapted (scotopic) testing done with the OCD, left eye followed by right eye. The non-tested eye may be covered during testing. After scotopic testing, the light of the OCD will be increased and light-adapted (photopic) testing will be performed in the same manner. 6) Debriefing. Subjective assessments of the testing modality and dark adaptation process will be collected.

*************************

Study 2: Study subjects participating in this portion of the study will require two study visits.

Potential participants will be approached by the PI to ask if they are willing to participate in this study. If the subject agrees to participate, during their next scheduled clinic visit, the PI will also do a slit lamp examination including lens status using the AREDS 2008 Clinical Lens Opacity Grading Standards in addition to their standard of care clinic eye visit. The slit lamp examination including lens status using the AREDS 2008 Clinical Lens Opacity Grading Standards is the only research related activity in this clinic visit. Potential participants who are the "normals" for Study 2 will be recruited from one of the co-investigator's clinic who is their treating physician. If interested, their physician (co-investigator) will contact the research coordinator to meet or call the patient and explain the study. If he/she agrees to participate, the PI will do a slit lamp examination at their next scheduled visit in the same manner as the other Study 2 participants, except the central corneal thickness will also be determined by ultrasonic pachymetry (standard testing for patients with glaucoma but not normal controls). Data from these clinic visits will be used as baseline information for the study. The baseline clinical and demographic data to be collected in the study will be: 1. Date of Birth 2. Ethnicity 3. Gender 4. Ocular History (surgery, etc) 5. Type of Glaucoma 6. Current visual acuity 7. Refraction 8. Central corneal thickness 9. Intraocular Pressure 10. Slit lamp examination including lens status by methods above 11. Dilated examination including optic nerve appearance 12. Recent automated perimetry results (Humphrey visual field)

Research Study Visit 1 (within 2 months of clinic visit from which clinical data is obtained):

1. Humphrey standard automated perimetry (visual field testing). This is a form of static perimetry used to assess retinal function and sensitivity. It is a commonly used photopic testing modality for the diagnosis and status of glaucoma and used frequently throughout ophthalmology and many ophthalmologic clinical studies. We hypothesize that there will be similarities in performance between Humphrey automated perimetry and OKR testing which will help validate our testing strategy. For patients with glaucoma, for whom visual field testing is frequently performed, this test will not be performed if a high-quality visual field test has been obtained within the last 6 months. For such patients, the visual field test from the clinical record will be used in the study.
2. OKR-based contrast testing will be performed with the OCD - optokinetic contrast device (the device in study with this protocol). Subjects will be shown a brief demonstration of the OCD under infrared light (to begin dark adaptation) to familiarize themselves with the device and the expected testing strategy.
3. Subjects will then be dark adapted for 20-30 minutes. During this time they may be blindfolded (depending on darkness of the room) and sitting in a dark room. Music options will be available to help pass the time and ease potential discomfort.
4. After 20-30 minutes, the blindfold will be removed (if used) and patient will have monocular dark-adapted (scotopic) testing done with the OCD, left eye followed by right eye. The non-tested eye may be covered during testing.
5. After scotopic testing, the light of the OCD will be increased and light-adapted (photopic) testing will be performed in the same manner.

This visit should take approximately 90 minutes to complete.

Second Research Visit (approximately 1 month after the first research visit):

1. Pelli-Robson Contrast Sensitivity Testing. This is a form of stationary central vision contrast sensitivity that is a commonly used testing modality for photopic contrast in many ophthalmologic clinical studies. We hypothesize that there will be similarities in contrast performance between Pelli-Robson and OKR testing which will help validate our testing strategy.
2. OKR-based contrast testing. This will be performed as in the second visit described above except that the testing order will be the right eye first, followed by the left eye.
3. Debriefing. Subjective assessments of the testing modality and dark adaptation process will be collected.

This visit should take approximately 90 minutes to complete.

For those participating in Study 2, participants will be asked if they will allow the study staff to review their medical records to track clinical outcomes for 5 years. Participants will be asked to allow review of their medical records related to their developing or not developing glaucoma or other eye conditions to collect longitudinal data. This is an optional portion of the test for which they can opt out.

The following information will be re-reviewed: 1. Date of Birth 2. Ethnicity 3. Gender 4. Ocular History (surgery, etc) 5. Type of Glaucoma 6. Visual acuity 7. Refraction 8. Central corneal thickness 9. Intraocular Pressure 10. Slit lamp examinations including lens status 11. Dilated examinations including optic nerve appearance 12. Automated perimetry results (Humphrey visual field)

ELIGIBILITY:
Inclusion Criteria:

Normal controls for Study 1

1. Male or Female
2. age 18 or older
3. Corrected visual acuity 20/40 or better in both eyes.

Normal Controls for Study 2

1. Male or Female
2. age 50 or older
3. IOP (intraocular pressure) 21 or less in both eyes
4. Corrected visual acuity 20/40 or better in both eyes.

Subjects with glaucoma/ocular hypertension

1. Male or Female
2. Age 50 or older
3. Defined as IOP> 21 without medication on two or more clinic visits in one or both eyes
4. Corrected visual acuity 20/40 or better
5. Normal optic nerves
6. Normal automated perimetry in both eyes

Subjects who are glaucoma/glaucoma suspects

1. Male or Female
2. Age 50 or over
3. Increased optic nerve cupping in one or both eyes regardless of IOP
4. Corrected visual acuity 20/40 or better
5. Normal automated perimetry in both eyes

Subjects with early to moderate glaucoma

1. Male or female
2. Age 50 or over
3. Increased optic nerve cupping regardless of IOP in one or both eyes
4. Corrected visual acuity 20/40 or better in both eyes
5. Early to moderate perimetric changes defined as a mean deviation (MD) no less than -7.5 and a pattern standard deviation (PSD) no greater than +7.5 in the worse eye.

Subjects with moderate to advanced glaucoma

1. Male of Female
2. Age 50 or older
3. Increased optic nerve cupping regardless of IOP in one or both eyes
4. Grossly abnormal automated perimetry (MD less than -7.5 or PSD greater than +7.5 in the worse eye)
5. Best-corrected visual acuity of 20/40 or better in both eyes

Exclusion Criteria:

* Normal Controls (both studies):

  1. glaucoma or glaucoma suspicion in either eye
  2. IOP > 21 in either eye
  3. History of use of IOP-reducing drops in either eye except temporarily following cataract extraction
  4. History of any ocular surgery except cataract extraction or refractive surgery (LASIK, PRK, or equivalent) in either eye
  5. Retinal disease in either eye
  6. Abnormal measured automated perimetry in either eye
  7. Abnormal measured contrast sensitivity in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J. Frankfort, M.D. PhD., Principal Investigator — Baylor College of Medicine
Locations (1):
- Alkek Eye Center, Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal subjects were recruited by word of mouth (medical clinic staff, employees, friends, relatives); Glaucoma subjects were recruited from a glaucoma specific clinic.
Units Other Than Participants: Eyes
Groups:
- Normal: Normal subjects without glaucoma
- Glaucoma: Subjects with glaucoma
Period: Overall Study
Arm/Group | Normal | Glaucoma
Started | 12; 24 Eyes | 11; 22 Eyes
Completed | 10; 20 Eyes | 10; 20 Eyes
Not Completed | 2; 4 Eyes | 1; 2 Eyes
Not completed — Unable to record log contrast sensitivity | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal | Glaucoma | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 5 | 17
  >=65 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
Best Corrected Vision = 20/40 or better [Count of Participants; unit: Participants] | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Estimated Contrast Sensitivity in Log Units (logCS)
Description: The HOCD willl be used to estimate the logCS of both eyes in both dark (scotopic) and light (photopic) conditions.
Time Frame: Study 1: Measured on the day of enrollment - reported only for those enrolled (early Termination). Study 2: Measured on the day of enrollment and 1 month later - not started (early Termination).
Population: Scotopic and photopic logCS for both eyes (right and left)
Measure: Median (Inter-Quartile Range); unit: logCS
Units Other Than Participants: Eyes
Arm/Group | Normal | Glaucoma
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 20 | 20
logCS
  Scotopic - right eyes: number analyzed (Eyes) | 10 | 10
  Scotopic - right eyes | 1.26 [1.19 to 1.58] | 1.50 [1.43 to 1.60]
  Scotopic - left eyes: number analyzed (Eyes) | 10 | 10
  Scotopic - left eyes | 1.45 [1.32 to 1.64] | 1.70 [1.35 to 1.91]
  Photopic - right eyes: number analyzed (Eyes) | 10 | 10
  Photopic - right eyes | 0.264 [-0.428 to 1.57] | -0.188 [-0.44 to 0.0417]
  Photopic - left eyes: number analyzed (Eyes) | 10 | 10
  Photopic - left eyes | 1.06 [-0.0663 to 1.62] | -0.0933 [-0.502 to 0.857]

2. Secondary Outcome: Compare Log Contrast Sensitivity in Subjects With and Without Glaucoma
Description: Measure differences in logCS between subjects with and without glaucoma.
Time Frame: as for outcome 1
Population: Scotopic and photopic logCS (right and left eyes pooled together)
Measure: Median (Inter-Quartile Range); unit: logCS
Units Other Than Participants: Eyes
Arm/Group | Normal | Glaucoma
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 20 | 20
logCS
  Scotopic - all eyes | 1.42 [1.22 to 1.58] | 1.52 [1.36 to 1.81]
  Photopic - all eyes | 0.65 [-0.322 to 1.59] | -0.188 [-0.462 to 0.536]
Statistical Analysis 1: Comparison: Normal vs Glaucoma; Test type: Other; p = 0.0583, Kruskal-Wallis — Scotopic logCS
Statistical Analysis 2: Comparison: Normal vs Glaucoma; Test type: Other; p = 0.1762, Kruskal-Wallis — Photopic logCS

3. Secondary Outcome: Compare Log Contrast Sensitivity Measured With the HOCD to White on White Sensitivity Via Automated Perimetry
Description: Measure contrast sensitivity with the HOCD (logCS) and then compare to automated perimetry results (Decibels). For subjects with glaucoma this will be performed as part of both Study 1 and Study 2. For normal control subjects, this will only be performed as part of Study 2.
Time Frame: Study 1: Measured on the day of enrollment - reported only for those enrolled (early Termination). Study 2: Measured on the day of enrollment - not started (early Termination).
Population: Only subjects with glaucoma had automated perimetry for comparison in Study 1. Eyes were pooled for analysis.
Measure: Mean (Standard Deviation); unit: Decibels
Units Other Than Participants: Eyes
Arm/Group | Normal | Glaucoma
Number analyzed (Participants) | 0 | 10
Number analyzed (Eyes) | 0 | 20
Decibels
  MD |  | -2.82 (3.27)
  PSD |  | 4.34 (3.41)
Statistical Analysis 1: Comparison: Glaucoma; Correlation between logCS and MD; Test type: Other; p = 0.183, Pearson correlation — Scotopic
Statistical Analysis 2: Comparison: Glaucoma; Correlation between logCS and MD; Test type: Other; p = 0.771, Pearson correlation — Photopic
Statistical Analysis 3: Comparison: Glaucoma; Correlation between logCS and PSD; Test type: Other; p = 0.492, Pearson correlation — Scotopic
Statistical Analysis 4: Comparison: Glaucoma; Correlation between logCS and PSD; Test type: Other; p = 0.830, Pearson correlation — Photopic

4. Secondary Outcome: Compare Contrast Sensitivity Measured With the HOCD to Contrast Sensitivity Testing Via Pelli Robson Contrast Sensitivity Chart Testing.
Description: Compare contrast sensitivity measured with the HOCD (logCS) to contrast sensitivity testing via Pelli Robson Contrast Sensitivity Chart testing. Study 2 only.
Time Frame: Study 2: Measured 1 month after the day of enrollment - not started (early Termination).
Population: Study 2 never performed due to early Termination
Arm/Group | Normal | Glaucoma
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Tolerance of Testing as Measured Via Questionnaire
Description: Subjects will be asked to relate their experiences with the test to determine how well it is tolerated. Subjects will be asked to report their agreement with five statements.
  This is reported on a custom scale: 1 = Do Not Agree; 2 = Partially Agree; 3 = Mostly Agree; 4 = Fully Agree.
  Higher scores represent more complete agreement with the statement.
Time Frame: Study 1: Measured on the day of enrollment - reported only for those enrolled (early Termination). Study 2: Measured 1 month after the day of enrollment - not started (early Termination).
Population: Only the subjects for whom testing was completed are described.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Normal | Glaucoma
Number analyzed (Participants) | 10 | 10
score on a scale
  I understood the test instructions. | 3.9 [3 to 4] | 4 [4 to 4]
  I was physically comfortable during the test. | 3.7 [3 to 4] | 3.6 [2 to 4]
  The length of the test was appropriate. | 2.8 [1 to 4] | 3.6 [2 to 4]
  I had problems with the time spent in the dark. | 1.3 [1 to 3] | 1 [1 to 1]
  I would recommend this test if likely to diagnose glaucoma sooner. | 4 [3 to 4] | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: Day of study enrollment
Description: Adverse events were monitored on the day of study enrollment. There were no return study dates.
Arm/Group | Normal | Glaucoma
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT02014597/Prot_SAP_000.pdf